CLINICAL TRIAL: NCT05163990
Title: Based on Non-invasive Cardiac Output Monitoring System to Explore the Preventive and Therapeutic Effect of Transcutaneous Acupoint Electrical Stimulation on Hypotension After Intraspinal Anesthesia in Cesarean Section
Brief Title: Study the Effect of Electroacupuncture on Prevention and Treatment of Hypotension After Intraspinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XJTU1AF2021LSK-332
Record Dates: First submitted 2021-11-10; First posted 2021-12-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-10

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: TEAS group: 10 minutes before intraspinal anesthesia, bilateral Neiguan points and Zusanli points are given dense wave transcutaneous acupoint electrical stimulation with the frequency of 10/50Hz. The intensity is based on the maximum tolerance of the participant, and the stimulation last until 30 minutes after subarachnoid administration.
  Control group: Electrodes are connected at bilateral Neiguan points and Zusanli points 10 minutes before intraspinal anesthesia, but no transcutaneous acupoint electrical stimulation is given, the duration is the same as that of the TEAS group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS group (Experimental): 10 minutes before intraspinal anesthesia, bilateral Neiguan points and Zusanli points are given dense wave transcutaneous acupoint electrical stimulation with the frequency of 10/50Hz. The intensity is based on the maximum tolerance of the participant, and the stimulation last until 30 minutes after subarachnoid administration.
  Interventions: Other: transcutaneous acupoint electrical stimulation
- Control group (No Intervention): Electrodes are connected at bilateral Neiguan points and Zusanli points 10 minutes before intraspinal anesthesia, but no transcutaneous acupoint electrical stimulation is given, the duration is the same as that of the TEAS group.

INTERVENTIONS:
Other: transcutaneous acupoint electrical stimulation — The corresponding transcutaneous acupoint electrical stimulation is given to different groups before spinal anesthesia, which last from 10 minutes before anesthesia to 30 minutes after subarachnoid administration.
  Arms: TEAS group

SUMMARY:
The purpose of this study is to assess the prevention and treatment effect of transcutaneous acupoint electrical stimulation on hypotension after intraspinal anesthesia.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo the doctors' and researchers' examination to determine eligibility for study entry. At beginning of the study, patients who meet the eligibility requirements will be randomized in a open manner（participant and electroacupuncture executor）in a 1:1 ratio to TEAS group (10 minutes before intraspinal anesthesia, bilateral Neiguan points and Zusanli points are given dense wave transcutaneous acupoint electrical stimulation with the frequency of 10/50Hz. The intensity is based on the maximum tolerance of the participant, and the stimulation last until 30 minutes after subarachnoid administration) or Control group (Electrodes are connected at bilateral Neiguan points and Zusanli points 10 minutes before intraspinal anesthesia, but no transcutaneous acupoint electrical stimulation is given, the duration is the same as that of the TEAS group).

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age < 55 years
* ASA classification I ~ II
* full term (37 weeks ≤ gestational weeks < 42 weeks)
* fchedule for elective single cesarean section under spinal anesthesia
* no other clinical trial 3 months before the enrollment
* volunteer to participate and sign the informed consent form

Exclusion Criteria:

* severe preeclampsia or hypertension
* diabetes
* cardiac insufficiency
* mental abnormality or cognitive impairment or inability to communicate
* acupuncture points skin breakage, infection, allergy
* the researchers believe that there are any conditions that are not suitable for inclusion.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
incidence of hypotension | within 30 minutes after subarachnoid administration
  the incidence of hypotension within 30 minutes after subarachnoid administration in TEAS group was significantly lower than that in Control group.

SECONDARY OUTCOMES:
specific changes of hemodynamic indexes | within 30 minutes after subarachnoid administration
  compared with Control group, the changes of hemodynamic indexes in TEAS group were more stable.
usage of ephedrine | within 30 minutes after subarachnoid administration
  the usage of ephedrine within 30 minutes after subarachnoid administration in TEAS group was significantly less than that in Control group.
incidence of nausea and vomiting | within 30 minutes after subarachnoid administration
  the incidence of nausea and vomiting within 30 minutes after subarachnoid administration in TEAS group was significantly lower than that in Control group.
incidence of dizziness, chest tightness and dyspnea | within 30 minutes after subarachnoid administration
  the incidence of dizziness, chest tightness and dyspnea within 30 minutes after subarachnoid administration in TEAS group was significantly lower than that in Control group.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, doctor, Study Chair — First Affiliated Hospital of Xian Jiaotong University; Ying Xiao, doctor, Study Director — First Affiliated Hospital of Xian Jiaotong University; Juan Bai, doctor, Study Director — First Affiliated Hospital of Xian Jiaotong University; Meng Yue Xu, postgraduate, Principal Investigator — Shaanxi University of Chinese Medicine
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arai YC, Kato N, Matsura M, Ito H, Kandatsu N, Kurokawa S, Mizutani M, Shibata Y, Komatsu T. Transcutaneous electrical nerve stimulation at the PC-5 and PC-6 acupoints reduced the severity of hypotension after spinal anaesthesia in patients undergoing Caesarean section. Br J Anaesth. 2008 Jan;100(1):78-81. doi: 10.1093/bja/aem306. Epub 2007 Oct 24. PMID 17959591

DOCUMENTS (2):
  • Study Protocol (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT05163990/Prot_000.pdf
  • Informed Consent Form (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT05163990/ICF_001.pdf